CLINICAL TRIAL: NCT03621826
Title: DISPLACE: Dissemination and Implementation of Stroke Prevention Looking at the Care Environment (Part 1 and 2)
Brief Title: Evaluating Barriers to Stroke Screening and Prevention in Children With Sickle Cell Disease
Acronym: DISPLACE
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00073134; R01HL133896 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-08-09 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Stroke Ischemic; Sickle Cell Disease
Keywords: sickle cell anemia; TCD; screening; dissemination; implementation
MeSH Terms: conditions — Ischemic Stroke; Anemia, Sickle Cell | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Sickle Cell Anemia: Data from patients with sickle cell anemia will be entered into a retrospective database for evaluation of implementation rates of TCD (stroke) screening). A small number of these children/parents/stakeholders will be selected by convenience sampling to participate in a survey and/or interview to assess barriers and enablers to stroke prevention therapy.
  Interventions: Other: Questionnaire/Interview

INTERVENTIONS:
Other: Questionnaire/Interview — A convenience sample of patients/parents and stakeholders will be asked to participate in a survey and/or interview to evaluate barriers to care in sickle cell.

SUMMARY:
DISPLACE is a three part, multi-center U.S. based study to evaluate the barriers to stroke screening and prevention in children with sickle cell anemia (SCA). In the United States, TCD (Transcranial Doppler ultrasound) is a proven method of screening children with SCA for stroke. However, many children are not getting the screening they need. This study will examine the issues that hinder and help children get the screening at 28 different hospitals and sickle cell centers to improve care for all children with sickle cell anemia. The investigators will then plan a study (part 3) aimed to improve stroke screening and prevention in sickle cell anemia.

DETAILED DESCRIPTION:
DISPLACE (Dissemination and Implementation of Stroke Prevention: Looking At the Care Environment) is a multi-center, national NHLBI-funded grant to evaluate the real world implementation of the STOP protocol in which transcranial Doppler (TCD), a measure of cerebral blood vessel velocity, is used to screen for stroke risk in children ages 2-16 with sickle cell anemia (SCA). Based on the STOP (Stroke Prevention Trial in Sickle Cell Anemia) protocol, children identified as high risk of stroke by TCD are initiated on chronic red cell transfusion therapy (CRCT) for stroke prevention. Children with normal TCD are screened annually from the age of 2 until they are 16 years of age.

This will be a THREE-part study beginning with Part 1 - a retrospective case record review followed by Part 2 - a multi-level qualitative assessment of barriers and enablers to TCD screening and initiation of chronic red blood cell transfusions and later adding Part 3 - a multi-center implementation clinical trial.The investigators will compare two implementation interventions to improve TCD screening.

There are three aims of the grant and each aim is equivalent to the respective parts of the grant (i.e. Part 1 covers 1 aim). There are a total 28 consortium sites. The Medical University of South Carolina is the lead institution for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age is >2 and <16 at time of review (from 2012-2016)
* have documented sickle cell anemia
* primary language is English
* patient at a DISPLACE consortium institution

Caregiver Characteristics:

Parent or guardian of patient who meets above criteria Primary language is English Has the cognitive capacity to complete questionnaires

EXCLUSION CRITERIA:

Child Characteristics:

Experiencing current acute complications of sickle cell disease requiring hospitalization or an acute care visit (e.g., pain crises, acute chest syndrome, acute cerebrovascular events/stroke or active infection/fever)

Caregiver Characteristics:

Has a child experiencing current acute complication of sickle cell disease, such as pain crisis, acute chest syndrome, stroke, or infection.

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with sickle cell anemia who were between 2-16 years of age from 2012-2016.
Sampling Method: Non-Probability Sample
Enrollment: 5247 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Annual TCD screening rates (retrospective data assessment) | 2 years
  Current rate of TCD screening over the last 5 years
Identify the barriers and enablers to TCD screening | 2 years
  This study will assess two different implementation strategies to improve TCD screening. To determine which strategy is more effective, a difference in TCD screening rates of at least 17% between intervention arms is necessary. If there is not at least a 17% difference in annual TCD screening rates, it will be impossible to determine the optimal implementation procedures
Retrospective assessment of initiation of chronic transfusion therapy in patients over the last 5 years in those children at risk of stroke | 2 years
  Patients with abnormal TCD should be started on chronic transfusion therapy. The goal of the intervention is to increase institutional initiation of CRCT in at least 95% of patients noted to have abnormal TCD

SECONDARY OUTCOMES:
Evaluate patient and stakeholder reported barriers to CRCT | 2 years
  The investigators will asses barriers to CRCT

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kanter, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No